CLINICAL TRIAL: NCT01326728
Title: Study of the Biology and Natural History of Disease Outcomes in Patients Treated With Allogeneic Hematopoietic Stem Cell Transplantation for Hematologic Malignancies
Brief Title: Relapsed Malignant Blood Cancer After Allogeneic Hematopoietic Stem Cell Transplantation
Status: Terminated | Type: Observational
Why Stopped: A replacement protocol was created to replace this current version of protocol.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ronald Gress, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110125; 11-C-0125
Record Dates: First submitted 2011-03-30; First posted 2011-03-31 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Chronic Myelogenous Leukemia; Acute Myelogenous Leukemia; Acute Lymphoblastic Leukemia; Hodgkins Lymphoma; Non-Hodgkins Lymphoma
Keywords: Relapse; Hematologic Malignancy; Allogeneic; Hematopoietic Stem Cell Transplantation; Leukemia; Lymphoma; Hodgkin Lymphoma
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin; Recurrence; Hematologic Neoplasms; Leukemia; Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue specimens collected in the course of this research project may be cryopreserved and used in the future to investigate new scientific questions related to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Allogeneic Stem Cell Transplant: Allogeneic hematopoietic stem cell transplantation (or allotransplant; donor blood stem cells)
  Interventions: Biological: Allogeneic stem cell transplant

INTERVENTIONS:
Biological: Allogeneic stem cell transplant — Donors will undergo cell collection and recipients will receive cells (allotransplant).

SUMMARY:
Background:

Allogeneic hematopoietic stem cell transplantation (or allotransplant; donor blood stem cells) have been used with varying degrees of success as an immune therapy for blood-system cancers (leukemias, myelodysplastic syndrome, lymphomas, multiple myeloma, etc.). Some people s cancer remains active (comes back or continues to spread) after an allotransplant, while other peoples cancer disappears and they are hopefully cured. National Institutes of Health (NIH) researchers are studying the reasons for these different treatment outcomes, and trying to develop better cancer treatments for people with active cancer after allotransplant. Researchers are collecting data from people who have had allotransplants for a cancer of the blood, whether or not the cancer is in remission, and from their donors. Those with active cancers may be eligible to participate in one of several NIH studies testing treatments for active cancer after allotransplant.

Objectives:

* To develop a systematic, comprehensive evaluation of individuals with relapsed malignant blood cancers after allotransplant (and, if available, their donors) to identify potential treatment study options
* To compare the immune system after allotransplant between people whose cancers are growing with people whose cancers remain in remission.
* To compare the immune system after cancer relapse/progression treatment between people whose cancer responds to treatment with those whose cancers continue to grow.

Eligibility:

* Individuals whose blood system cancer grows or comes back after receiving allotransplant treatment.
* Individuals whose blood system cancer is responding or in remission 100 days or more after receiving allotransplant treatment.
* Related stem-cell donors of eligible allotransplant recipients.

Design:

* Participants will be evaluated with a full physical examination, detailed medical history (for recipients, including a history of allotransplant treatment process, side-effects, etc.), and blood tests. Recipients will also have imaging studies, possible tissue biopsies, quality of life questionnaires/assessments, and other tests to evaluate the current state of their cancer, whether active or in remission. In some cases, it may be possible to substitute results from recent tests and/or biopsies.
* Healthy related donors will have apheresis to provide white blood cells for study and/or for use in potential treatment options. If stem cells would be medically helpful to a recipient, their donors might be asked to take injections of filgrastim before the apheresis procedure to stimulate the production of stem cells for collection.
* As feasible, all recipients will be asked to return to the NIH for detailed follow-up visits in conjunction with 6, 12, and 24 months post-allotransplant evaluations, and may be monitored between visits.
* Recipients whose cancers are active and who are found to be eligible for treatment protocols at the NIH will continue to be monitored on this study while participating on treatment protocols. Return visits and follow-up tests for this study will be coordinated with those required by the treatment protocol.
* Participants may return in the future to be evaluated for new treatment study options (recipients) or additional cell donations for therapy (donors).

DETAILED DESCRIPTION:
Background:

* Cancer relapse is a significant clinical problem following allogeneic hematopoietic stem cell transplantation (allotransplant), affecting up to half of all patients. Effective treatment options are extremely limited and, for most cancers, rarely curative.
* Several Clinical Center (CC) protocols are evaluating treatment for post-allotransplant relapse. Relapse often progresses quickly; patients require rapid assessment of protocol options in order to expedite initiation of treatment.
* Basic information is needed to improve management of relapse after allotransplant clinical information regarding risk of relapse and cancer behavior after allotransplant, and information on the biology of relapse after allotransplant in order to identify risk factors, target prevention strategies, detect early relapse and develop effective treatments.

Objectives:

Primary Objective:

To provide a mechanism for systematic, comprehensive evaluation of individuals with relapsed hematologic malignancy after allotransplant and, if available, their donors, to streamline identification of protocol options, enrollment and initiation of therapy.

Eligibility:

1. Individuals who have received allotransplant treatment for hematologic malignancy ("Recipient-Subjects"). Analyses (secondary aims) will consider two comparison cohorts:

   1. Relapse Cohort: Cancer progression, relapse or persistently stable (unremitting) disease
   2. Remission (Control) Cohort: Cancer response or remission at/after Day 100
2. Individuals who are being enrolled on Clinical Center protocols to undergo allotransplant therapy for hematologic malignancies and are being evaluated at the Clinical Center for planned allotransplantation. (Recipient-Subjects)
3. Related donors of eligible allotransplant recipients ("Donor-Subjects")

Design:

1. Recipient-Subjects will have clinical and research evaluations at baseline and three and six months post-allotransplant, at six-month intervals through three years post-allotransplant, then yearly. Evaluation after relapse treatment response and for new protocol options is permitted.
2. Donor-Subjects will be enrolled at the time of their clinical evaluation and cell collection for Recipient-Subject therapy. Return evaluation for additional clinical product collection is permitted.
3. Accrual Ceiling: 500 consented subjects (350 Recipient-Subjects and 150 Donor-Subjects) over 5 years, averaging 70 Recipient-Subjects and 30 Donor-Subjects enrolled per year.

ELIGIBILITY:
* INCLUSION CRITERIA:

RECIPIENT SUBJECTS:

1. Individuals who are candidates for allotransplant therapy for hematologic malignancies and are being evaluated at the Clinical Center for planned allotransplantation.
2. Individuals who have received allotransplant treatment for hematologic malignancy and have:

   1. Hematologic recovery after allotransplant: e.g., have had neutrophil recovery to 500 cells/mcL. Secondary cytopenias or cytopenias due to disease progression will be permitted. Note: this requirement will not apply to subjects enrolling pre-transplant, i.e, who receive transplant-related medical care at the Clinical Center (CC).
   2. An ongoing relationship with a primary oncologist who will continue to provide continuity of care during and after study participation.
   3. Following record review and information exchange between the patients primary oncologist and the National Cancer Institute (NCI) Principal Investigator (PI)/Designee, the PI/Designee determines that the individual reasonably could be expected to safely tolerate travel to and from the Clinical Center (CC) to undergo evaluation as defined in the protocol, in the event that the patient is ineligible or uninterested in participating in open treatment protocols.
3. 18-99 years.
4. Ability of subject to understand and the willingness to sign a written informed consent document.

DONOR SUBJECTS:

1. Individuals who are/will be the donors of allogeneic hematopoietic stem cell transplants received by Recipient-Subjects who are to be enrolled on this protocol.
2. Age 18-99 years.
3. Ability of the subject to understand and the willingness to sign a written informed consent document.
4. Individuals with evidence of infection with transfusion-transmittable agents (Hepatitis B and C Viruses (HBV, HCV); Human Immunodeficiency Virus (HIV (Omega)), Human TLymphotrophic Virus (HTLV I/II), West Nile Virus (WNV) and Trypanosoma cruzi) will not be excluded from study participation. However, Donor-Subjects with evidence of HIV infection will only be able to donate cells for research. Donors with a history of HBV or HCV infection will be able to donate for research, and may be eligible to donate for therapeutic administration. However, determination of permissibility for clinical donation will require a hepatology consultation and the consent of the intended recipient after discussion of the risk/benefit of the donor cell product and the possibility/consequences of transmission. The PI/Designee will make the final determination of permissibility of donation for recipient cell therapy.

6. Unrelated donor selection will be in accordance with the National Marrow Donor Program (NMDP) standards. When a potentially eligible recipient of an unrelated donor product from an NMDP Center is identified, the recipient will complete an NMDP search transfer request to allow NIH NMDP staff to contact the NMDP Coordinating Center, who will, in turn, contact the donors prior Donor Center. The NMDP Policy for Subsequent Donation Requests will be followed and the appropriate forms (Subsequent Donation Request Form and Therapeutic T Cell Collection Prescription Form) will be submitted as required.

EXCLUSION CRITERIA:

RECIPIENT SUBJECTS:

1. Individuals with rapid disease progression or aggressive cancer histology who, in the opinion of the PI/Designee, require urgent therapy within 30 days in order to preserve organ function or quality of life. This restriction will not apply if there is no approved therapy with a reasonable chance of disease response, if the patient does not have access to an effective therapy and the patient appears to be eligible for an accruing CC treatment protocol or if the patient is enrolled on an NIH/CC clinical protocol, e.g., allotransplant protocol.
2. Pregnancy or lactating. Additionally, Recipient-Subjects of childbearing potential that will receive cancer treatment under this protocol must be willing to use an effective method of contraception.

DONOR SUBJECTS:

1. Adult donors who are not eligible for clinical donation will not be excluded from study participation, but will only be able to donate cells for research.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals aged 18-99 who are being enrolled on Clinical Center protocols to undergo allotransplant therapy for hematologic malignancies. The population will consist of those that have received allotransplant treatment for hematologic malignancy, are in remission either at or after Day 100, have malignancy progression or persistently stable disease post allotransplant, or the related donor of eligible allotransplant recipients.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2011-03-30 (Actual); Primary Completion 2017-06-28 (Actual); Study Completion 2017-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald E Gress, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pavletic SZ, Kumar S, Mohty M, de Lima M, Foran JM, Pasquini M, Zhang MJ, Giralt S, Bishop MR, Weisdorf D. NCI First International Workshop on the Biology, Prevention, and Treatment of Relapse after Allogeneic Hematopoietic Stem Cell Transplantation: report from the Committee on the Epidemiology and Natural History of Relapse following Allogeneic Cell Transplantation. Biol Blood Marrow Transplant. 2010 Jul;16(7):871-90. doi: 10.1016/j.bbmt.2010.04.004. Epub 2010 Apr 24. PMID 20399876
- [Background] Dazzi F, Fozza C. Disease relapse after haematopoietic stem cell transplantation: risk factors and treatment. Best Pract Res Clin Haematol. 2007 Jun;20(2):311-27. doi: 10.1016/j.beha.2006.10.002. PMID 17448964
- [Background] Porter DL, Alyea EP, Antin JH, DeLima M, Estey E, Falkenburg JH, Hardy N, Kroeger N, Leis J, Levine J, Maloney DG, Peggs K, Rowe JM, Wayne AS, Giralt S, Bishop MR, van Besien K. NCI First International Workshop on the Biology, Prevention, and Treatment of Relapse after Allogeneic Hematopoietic Stem Cell Transplantation: Report from the Committee on Treatment of Relapse after Allogeneic Hematopoietic Stem Cell Transplantation. Biol Blood Marrow Transplant. 2010 Nov;16(11):1467-503. doi: 10.1016/j.bbmt.2010.08.001. Epub 2010 Aug 10. PMID 20699125

RESULTS

PARTICIPANT FLOW:
Groups:
- Recipients: Recipient-Subjects will have clinical and research evaluations at baseline and three and six months post-allotransplant, at six-month intervals through three years post-allotransplant, then yearly. Evaluation after relapse treatment response and for new protocol options is permitted.
- Donors: Donor-Subjects will be enrolled at the time of their clinical evaluation and cell collection for Recipient-Subject therapy. Return evaluation for additional clinical product collection is permitted.
Period: Overall Study
Arm/Group | Recipients | Donors
Started | 47 | 9
Completed | 0 | 0
Not Completed | 47 | 9
Not completed — Death | 13 | 0
Not completed — Early closure of study | 34 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Recipients | Donors | Total
Number analyzed (Participants) | 47 | 9 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 9 | 48
  >=65 years | 8 | 0 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.34 (15.46) | 50.33 (14.54) | 49.83 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 3 | 23
  Male | 27 | 6 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 40 | 8 | 48
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 38 | 5 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 47 | 9 | 56
Count of Participants with Presence or Absence of GVHD Prior to Study [Count of Participants; unit: Participants] — Recipients only (study specific baseline measure not applicable to donors) were assessed for graft versus host disease (GVHD) prior to study. GVHD is a medical complication following stem cell transplant that can affect the skin, gut, and various other parts of the body. Since the baseline would be pre-transplant, no patient would have GVHD and would have captured as a general patient assessment. Because this was a natural history study, this data may have come from a transplant that occurred before they were on study.
  Participants
    Presence of GVHD | 0 | NA — Healthy related donors underwent apheresis and provided white blood cells for study and/or for use in potential treatment options. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Absence of GVHD | 47 | NA — Healthy related donors underwent apheresis and provided white blood cells for study and/or for use in potential treatment options. | NA — Total not calculated because data are not available (NA) in one or more arms.
Count of Participants with Disease Present Prior to Stem Cell Transplant Conditioning [Count of Participants; unit: Participants] — Patients were receiving transplants to treat present disease of multiple varieties, so all patients would have had disease present at time of transplant. Because this was a natural history study, this data may have come from a transplant that occurred before they were on study.
  Participants | 47 | NA — Healthy related donors underwent apheresis and provided white blood cells for study and/or for use in potential treatment options. | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Immune Suppression
Description: Biological response to agents and or treatments that can lead to bone marrow suppression/ cytopenias and sometimes death.
Time Frame: up to 100 days or more following transplant
Population: Protocol specified data were not to be summarized or analyzed unless 30-40 total pts in both grps (no relapse, relapse) are available (to permit a given comparison to have approx. 80% power for a test with an effect size of 1.0 and 0.05 two-sided alpha level). PI of the study left the NIH before this number was reached and the study was terminated.
Arm/Group | Recipients
Number analyzed (Participants) | 0

2. Primary Outcome: Time to Progression After Allotransplant
Description: Time to Progression is the time between the first day of treatment to day 100 after allotransplant.
Time Frame: first day of treatment to day 100 after allotransplant
Population: as for outcome 1
Arm/Group | Recipients
Number analyzed (Participants) | 0

3. Primary Outcome: Overall Survival
Description: Overall Survival is the time between the first day of treatment to the day of death.
Time Frame: first day of treatment to the day of death
Population: as for outcome 1
Arm/Group | Recipients
Number analyzed (Participants) | 0

4. Primary Outcome: Days to Engraftment
Description: Number of days for a participant to reach engraftment.
Time Frame: up to 100 days or more following allotransplant
Population: as for outcome 1
Arm/Group | Recipients
Number analyzed (Participants) | 0

5. Primary Outcome: Count of Participants With Acute Graft Versus Host Disease (GVHD) Grade 2 or More 100 Days Post Allotransplant
Description: Acute GVHD is defined as GVHD that presents with signs and symptoms typical of acute GVHD but presenting after day 100 post allotransplant. Clinical Staging Grade 2 ((+) to (+++) Skin; (+) Liver; and (+) Gut) involvement, Grade 3 ((++) to (+++) Skin; (++ to +++) Liver; and (++ to +++) Gut) involvement, and Grade 4 ((++) to (++++) Skin; (++ to ++++) Liver; and (++ to ++++) Gut) involvement.
Time Frame: 100 days or more post allotransplant
Population: as for outcome 1
Arm/Group | Recipients
Number analyzed (Participants) | 0

6. Primary Outcome: Count of Participants With Chronic Graft Versus Host Disease (GVHD) Grade 2 or More 100 Days Post Allotransplant
Description: Mild chronic GVHD involves only 1 or 2 organs or sites with no clinically significant functional impairment (max. score of 1 in all affected organs or sites). Moderate GVHD involves at least 1 organ or site with clinically significant but no major disability (max. score of 2 in any affected organ or site), or 3 or more organs or sites with no clinically significant functional impairment (max. score of 1 in all affected organs or sites), and a lung score of 1 will also be considered moderate chronic GVHD. Severe chronic GVHD indicates major disability caused by chronic GVHD (score of 3 in any organ or site). A lung score of 2 or greater will also be considered severe chronic GVHD.
Time Frame: 100 days post allotransplant
Population: as for outcome 1
Arm/Group | Recipients
Number analyzed (Participants) | 0

7. Primary Outcome: Count of Participants With Infection After Allotransplant
Description: Count of Participants with Infection After Allotransplant.
Time Frame: up to 100 days or more post allotransplant
Population: as for outcome 1
Arm/Group | Recipients
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Recipients
Number analyzed (Participants) | 47
Participants | 13

9. Other Pre Specified Outcome: Count of Participants With Clinical Blood Markers of Inflammation
Description: Count of participants with clinical blood markers of inflammation. Normal to low blood markers indicate relapse. Falling blood marker levels indicate possible imminent relapse.
Time Frame: up to 100 days or more following allotransplant
Population: as for outcome 1
Arm/Group | Recipients
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: Regimen-Specific Sensitivity After Allotransplant
Description: Regimen-specific sensitivity are new or renewed sensitivity to therapies following allotransplant.
Time Frame: up to 100 days or more following allotransplant
Population: as for outcome 1
Arm/Group | Recipients
Number analyzed (Participants) | 0

11. Other Pre Specified Outcome: Tumor Immune Response Graft-Versus-Leukemia (GVL)
Description: GVL is a donor anti-tumor response following transplant.
Time Frame: up to 100 days or more following allotransplant
Population: as for outcome 1
Arm/Group | Recipients
Number analyzed (Participants) | 0

12. Other Pre Specified Outcome: Relapse After Day 100 or Following Treatment of Graft Versus Host Disease (GVHD)
Description: Participants who were initially in remission.
Time Frame: After Day 100 or Following Treatment of GVHD
Population: as for outcome 1
Arm/Group | Recipients
Number analyzed (Participants) | 0

13. Other Pre Specified Outcome: Recovery of Clinical Immunity After Allotransplant
Description: Improved serologic responses after allotransplant.
Time Frame: up to 100 days or more following allotransplant
Population: as for outcome 1
Arm/Group | Recipients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 5 years
Description: This protocol only captured grade 5 adverse events. it is a natural history study. All of the adverse events were captured on the subject's treatment/main protocol.
Arm/Group | Recipients | Donors
All-Cause Mortality (participants affected / at risk) | 13/47 | 0/9
Serious Adverse Events (participants affected / at risk) | 13/47 | 0/9
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recipients (N=47) | Donors (N=9)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Death
Sepsis (Infections and infestations) | 1 (1) | 0 (0) — Death
Treatment Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 0 (0) — Death

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-02-16): https://cdn.clinicaltrials.gov/large-docs/28/NCT01326728/Prot_SAP_ICF_000.pdf